CLINICAL TRIAL: NCT05682313
Title: Validity of Strain Elastography for the Evaluation of Chronic Allograft Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Associate professor, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD-53-2021
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Chronic Allograft Nephropathy
Keywords: Nephropathy, Chronic Tubulointerstitial; Kidney Transplantation; ultrasonography; Elasticity Imaging Techniques
MeSH Terms: conditions — Nephropathy, Chronic Tubulointerstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elastography arm (Experimental): single arm that includes all patient who have consented for ultrasound elastography
  Interventions: Diagnostic Test: Elastography arm

INTERVENTIONS:
Diagnostic Test: Elastography arm — Renal ultrasound elastography to detect and classify the degree of fibrosis

SUMMARY:
Chronic allograft nephropathy is one of dreaded complication of kidney transplant. It is one of the major determinants of long term graft survival. There are a number of factors that can contribute to chronic allograft nephropathy including chronic use of calcineurin inhibitors. Renal biopsy is the investigation of choice to detect chronic renal allograft nephropathy. renal biopsy has a number of complications . This includes infection and bleeding. The non invasive renal sono-elastography (strain and Shear Wave Imaging) technique has shown very good yield of detecting and scoring fibrosis.

In this study our aim is to determine the sensitivity and specificity of ( strain sono-elastography) in the detection and classifying of chronic allograft nephropathy as compared to transcutaneous renal biops

DETAILED DESCRIPTION:
Chronic allograft nephropathy is one of dreaded complication of kidney transplant. It is one of the major determinants of long term graft survival. There are a number of factors that can contribute to chronic allograft nephropathy including chronic use of calcineurin inhibitors. Renal biopsy is the investigation of choice to detect chronic renal allograft nephropathy. renal biopsy has a number of complications . This includes infection and bleeding. The non invasive renal sono-elastography (strain and Shear Wave Imaging) technique has shown very good yield of detecting and scoring fibrosis.

In this study our aim is to determine the sensitivity and specificity of ( strain sono-elastography) in the detection and classifying of chronic allograft nephropathy as compared to transcutaneous renal biopsy

ELIGIBILITY:
Inclusion Criteria:

Renal transplant patients of more than 2 years duration, Chronic allograft nephropathy proved by renal biopsy done within 1 month from the date of the strain elastography, Body mass index less than 30 kg/m2, Skin allograft distance of less than 3.5 cm, Parenchyma thickness of more than 1 cm and no fluid accumulation around the allograft.

Exclusion Criteria:

Body mass index more than 30 kg/m2, Skin allograft distance more than 3.5 cm, Parenchymal thickness less than 1 cm, Presence of any fluid collection around the allograft, GFR less than 15 ml/min, Graft stones or backpressure and less than 14 years old or more than 55 years old.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Grade of fibrosis | At the time of recruitment
  degree of fibrosis obtained by elastography

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelaziz, Principal Investigator — Kasr Alaini University Hsopitals
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No